CLINICAL TRIAL: NCT01274533
Title: A Phase II Study of Lenalidomide in Patients With Relapsed or Refractory HTLV-1 Associated Adult T Cell Leukemia/Lymphoma
Brief Title: Lenalidomide in HTLV-1 Adult T-Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAE5097
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Adult T Cell Leukemia/Lymphoma
Keywords: ATLL
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia-Lymphoma, Adult T-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Oral lenalidomide is initiated on Day 1 of Cycle 1 and continues once daily days 1-21 of a 28 day cycle. Subjects may continue participation in the Treatment Phase of the study for 24 months unless disease progression or drug is discontinued for safety reasons.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 25mg or 10mg (based on creatinine clearance) once daily for days 1-21 of a 28 day cycle
  Other Names: Revlimid

SUMMARY:
This is a research study for subjects who have been diagnosed with Adult T cell Leukemia/Lymphoma, a rare and aggressive peripheral T cell neoplasm caused by the virus HTLV1. Currently, there is no accepted standard therapy for this disease. The purpose of this research study is to evaluate the use of the investigational drug lenalidomide in the treatment of Adult T cell Leukemia/Lymphoma.

Lenalidomide is a drug that alters the immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may reduce or prevent the growth of cancer cells.

Lenalidomide is approved by the Food and Drug Administration (FDA) for the treatment of specific types of myelodysplastic syndrome (MDS) and in combination with dexamethasone for patients with multiple myeloma (MM) who have received at least 1 prior therapy. MDS and MM are cancers of the blood. It is currently being tested in a variety of cancer conditions. In this case it is considered experimental.

DETAILED DESCRIPTION:
The Primary Objective is to determine the efficacy of lenalidomide monotherapy in relapsed or refractory HTLV 1 associated Adult T Cell Leukemia/Lymphoma. Efficacy will be assessed by measuring the response rate, tumor control rate, duration of response, time to progression and progression free survival.

The Secondary Objective is to evaluate the safety of lenalidomide monotherapy as treatment for subjects with relapsed or refractory HTLV 1 associated Adult T Cell Leukemia/Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Relapsed or refractory HTLV-1 associated Adult T-cell Leukemia/Lymphoma (Acute and lymphoma subtypes)
* All previous cancer therapy, including radiation, hormonal therapy and surgery, must have been discontinued at least 4 weeks prior to treatment in this study.
* ECOG performance status of ≤ 2 at study entry (see Appendix C).
* Laboratory test results within these ranges:

  * Absolute neutrophil count ≥ 1000/mm³
  * Platelet count ≥ 50,000 /mm³
  * Calculated creatinine clearance of ≥ 30 mL/min by Cockcroft-Gault formula (Appendix J). Patients with calculated creatinine clearance ≥ 30 mL/min and < 60 mL/min will have a reduced starting dose of lenalidomide (see Section 5.4.2).
  * Total bilirubin ≤ 1.5 x ULN
  * AST (SGOT) and ALT (SGPT) ≤ 3 x ULN.
* Disease free of prior malignancies for ≥ 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix A: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods, AND also Appendix B: Education and Counseling Guidance Document.
* Patients at high risk for DVT/PE must be able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Evidence of laboratory TLS by Cairo-Bishop Definition of Tumor Lysis Syndrome (see Appendix H). Subjects may be enrolled upon correction of electrolyte abnormalities.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of lenalidomide.
* Concurrent use of other anti-cancer agents or treatments.
* Known positive for HIV or infectious hepatitis, type B or C.
* Recent DVT/PE requiring dose adjustments of anticoagulation within past 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-12; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne A Phillips, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in Aug. 2013.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 4
Completed | 0
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Non-compliance | 1
Not completed — Disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 4
Age, Customized [Number; unit: participants]
  18 years and older | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (CR + Cru + PR)
Description: Peripheral blood, CT or MRI
Time Frame: 28 days
Population: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in Aug. 2013.
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

2. Secondary Outcome: Safety of Lenalidomide Monotherapy
Time Frame: 28 days
Population: as for outcome 1
Arm/Group | Lenalidomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the AE data.
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No